CLINICAL TRIAL: NCT01824680
Title: Effect of a 3 Months Physical Activity Program on the Hormonal Regulation of Food Intake by Intense Physical Activity in Overweight Adolescents
Brief Title: Effect of a Physical Activity Program on the Hormonal Regulation of Food Intake
Acronym: APHRO
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0149
Record Dates: First submitted 2013-02-28; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: Obesity
Keywords: Obesity; Appetite regulation; Hormones; Adolescents; Exercise
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Exercise

ARMS (1):
- obesity (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — There is two sequences, one before and one after the physical activity program. Each sequence contains one "rest" session and one "exercise" session

SUMMARY:
The primary purpose of this protocol is to assess the hormonal regulation of satiety by an intense exercise before and after a 3 month physical activity program. Hormones assessed are: leptin, grhélin, Cholecystokinin, Glucagon-Like-Peptid-1 (GLP-1), PYY.

It is well known that in overweight adults and children also, an intense physical exercise diminish the food intake relatively to the total energy expenditure and this effect is persistent after a 6 weeks physical activity program.

Our hypothesis are: a diminution of food intake after the intense physical exercise and a persistent diminution of food intake after the 3 month physical activity program, an augmentation of levels of GLP-1 and PYY during the intense exercise before and after the physical activity program, a diminution of the level of GLP-1 and leptin before and after the physical activity program

DETAILED DESCRIPTION:
There is two sequences, one before and one after the physical activity program. Each sequence contains one "rest" session and one "exercise" session.

Each session contains : blood sample at regular interval (Leptin, Ghrélin, CCK, PYY, GLP-1), a sleeping assessment (Pittsburg scale), an assessment of hunger sensations at regular interval, an assessment of food intake in a "ad libitum" lunch and in the diner indirectly by the SU.VI.MAX. tool.

During the " rest " session :

Blood samples, assessment of hunger sensation, assessment of food intake are realized during the morning. Physical condition (VO2 max, DEXA, and muscular test), insulin-sensibility, lipid profile, are also assessed.

During the "exercise" session: it is identical to the first session but an intense exercise of 40 minutes is realized at 70% of the patient's VO2 max. The peripherical blood output is measured by a non-invasive method: the Near-Infra-Red-Spectroscopy, during the exercise.

The 3-months-physical activity program : there is 4 sessions of 30 minutes and 2 sessions of 1 hour per week. Most of exercises sessions are realized at home but one 1-hour session per week is controled with a sports educator.

ELIGIBILITY:
Inclusion Criteria:

Overweight adolescents (over the 90 th percentile of the international cut-off point)

* With a computer and an internet connection
* Sedentary (according to the IPAQ-A questionnaire)
* Without eating disorders (according to the DEBQ questionnaire)

Exclusion Criteria:

* Medical or surgical antecedents that are incompatible with the study: cardiovascular, endocrine or digestive disease.
* Drugs that could interfere with the results of the study
* Surgical intervention in the 3 months
* Regular consumption of tobacco or Alcohol
* patients on a diet with caloric restriction
* Refusal to sign the consent form
* Regular practice of sport and intensive

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-05 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Comparison before and after the physical activity program of the effect of intense exercise on kinetic of secretion of regulation hormones: Leptin, Grhélin, CCK, PYY3-36, GLP-1 | after 3 months of physical activity

SECONDARY OUTCOMES:
Comparison, before and after the physical activity program, of Hunger sensation by Visual Analogic Scales | after 3 months of physical activity
Comparison, before and after the physical activity program of food intake | after 3 months of physical activity
Comparison, before and after the physical activity program of insulinosensibility | after 3 months of physical activity
Comparison, before and after the physical activity program of peripheral blood output | after 3 months of physical activity
Comparison, before and after the physical activity program of sleep quality | agter 3 months of physical activity
Comparison, before and after the physical activity program of physical condition | after 3 months of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Etienne MERLIN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France